CLINICAL TRIAL: NCT05103098
Title: Sublingual Misoprostol 400 mcg and 800 mcg In Medical Treatment of First Trimester Missed Miscarriage: A Randomized Controlled Trial
Brief Title: Sublingual Misoprostol In Medical Treatment of First Trimester Missed Miscarriage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: hany farouk (Other)
Responsible Party: Sponsor-Investigator, hany farouk, Clinical Professor, Aswan University Hospital
Organization: Aswan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: aswu/354/9/19
Record Dates: First submitted 2021-10-14; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Miscarriage
Keywords: miscarriage; sublingual; misoprostol
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Misoprostol

STUDY DESIGN:
Intervention Model Description: a double-blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: a double-blind randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- misoprostol 400 mcg (Experimental): All patients will receive three doses of sublingual misoprostol every four hours The first dose of misoprostol 400 mcg will be administrated at the hospital. Then the patient will be observed for 1 hour for any immediate adverse reaction Clear instructions about the method and timing of the second dose will be given upon sending home.
  Two doses of misoprostol 800 mcg each (2 tablets of 200 mcg per dose). Paracetamol, eight hourly, will be provided as an analgesic or antipyretic. A specimen bottle to collect the POC if passed out. Two pairs of disposable gloves. Pre-filled histopathological examination form to be sent to the laboratory together with the products of conception
  Interventions: Drug: misoprostol 400 mcg
- misoprostol 800 mcg (Active Comparator): All patients will receive three doses of sublingual misoprostol every four hours The first dose of misoprostol 800 mcg will be administrated at the hospital. Then the patient will be observed for 1 hour for any immediate adverse reaction Clear instructions about the method and timing of the second dose will be given upon sending home.
  Two doses of misoprostol 800 mcg each (four tablets of 200 mcg per dose). Paracetamol, eight hourly, will be provided as an analgesic or antipyretic. A specimen bottle to collect the POC if passed out. Two pairs of disposable gloves. Pre-filled histopathological examination form to be sent to the laboratory together with the products of conception
  Interventions: Drug: misoprostol 800 mcg

INTERVENTIONS:
Drug: misoprostol 400 mcg — All patients will receive three doses of sublingual misoprostol every four hours The first dose of misoprostol 400 mcg will be administrated at the hospital. Then the patient will be observed for 1 hour for any immediate adverse reaction Clear instructions about the method and timing of the second dose will be given upon sending home.
  Two doses of misoprostol 400 mcg each (four tablets of 200 mcg per dose). Paracetamol, eight hourly, will be provided as an analgesic or antipyretic. A specimen bottle to collect the POC if passed out. Two pairs of disposable gloves. Pre-filled histopathological examination form to be sent to the laboratory together with the products of conception
  Other Names: experimental
  Arms: misoprostol 400 mcg
Drug: misoprostol 800 mcg — All patients will receive three doses of sublingual misoprostol every four hours The first dose of misoprostol 800 mcg will be administrated at the hospital. Then the patient will be observed for 1 hour for any immediate adverse reaction Clear instructions about the method and timing of the second dose will be given upon sending home.
  Two doses of misoprostol 800 mcg each (four tablets of 200 mcg per dose). Paracetamol, eight hourly, will be provided as an analgesic or antipyretic. A specimen bottle to collect the POC if passed out. Two pairs of disposable gloves. Pre-filled histopathological examination form to be sent to the laboratory together with the products of conception
  Other Names: Active Comparator
  Arms: misoprostol 800 mcg

SUMMARY:
The aim of this work is to compare the effectiveness of sublingual misoprostol 400 mcg versus 800 mcg for medical treatment of the first trimester missed miscarriage.

DETAILED DESCRIPTION:
the study will be made on female patients with the first trimester missed abortion confirmed by ultrasound. Participants will be divided into 2 groups one group (A) will receive sublingual Misoprostol 400 mcg and the other group(B) will receive sublingual Misoprostol 800 mcg every 4 hours in both groups up to 3 doses the aim of the study is to compare the efficacy of sublingual Misoprostol in complete termination of the first trimester missed abortion and which route is the best will less side effects.

ELIGIBILITY:
Inclusion Criteria:

* All women above 18 years of age
* Less than 12 weeks of gestation.
* Pregnancy is confirmed by pregnancy test or ultrasound scan.
* missed abortion
* Normal general and gynecological examination.

Exclusion Criteria:

* Hemodynamically unstable.
* Suspected sepsis with temperature 38 °C.
* Concurrent medical illness e.g. hematological, cardiovascular, thromboembolism,
* respiratory illnesses, recent liver disease, or pruritus of pregnancy.
* Presence of intrauterine contraceptive device (IUCD).
* Suspect or proven ectopic pregnancy.
* Failed medical or surgical evacuation before the presentation.
* Known allergy to misoprostol.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women with missed abortion in the first trimester
Enrollment: 200 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Completeness of abortion | 7 days
  Number of Participants with expulsion of Products of conception by visual inspection

SECONDARY OUTCOMES:
Successful medical abortion | 7 days
  Number of Participants with cervical os is closed with endometrial thickness of less than 15 mm
amount of calculated blood loss following treatment | 7 days
  amount of calculated blood loss

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No